CLINICAL TRIAL: NCT04151576
Title: The Effect of Aromatherapy Massage on the Pain Severity and Quality of Life in Acute Migraine Attacks
Brief Title: Aromatherapy Massage in Migraine Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Halic University (Other); Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Leman Şenturan, Prof. Dr., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Biruni U
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Pain; Head Pain; Quality of Life
Keywords: aromatherapy; massage
MeSH Terms: conditions — Pain; Headache

STUDY DESIGN:
Intervention Model Description: Randomized controlled experiment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The patients received medical treatment. The intervention: An aromatic oil mixture (lavender and peppermint) was massaged for 15 minutes on the temple and root of the neck of the patients, and this application continued for three weeks
  Interventions: Other: aromatherapy massage
- Control (No Intervention): The patients received only medical treatment

INTERVENTIONS:
Other: aromatherapy massage — aromatherapy massage
  Arms: Experimental

SUMMARY:
The aim of the study was to determine the effect of aromatherapy massage on the pain severity and quality of life in patients diagnosed with migraine in addition to medical treatment during an acute migraine attack.

In addition to medical treatments, complementary and supportive therapies are commonly used to cope with pain during a migraine attack. In recent years, aromatherapy through massage has become more common to reduce the severity of pain, make the patient painless and improve the quality of life. Aromatherapy applications are the application of pain relief oil mixtures through massage. Lavender and peppermint essential oils are mostly used in aromatherapy applications to reduce pain. Therefore, a mixture of mint and lavender oil was used in the study.

DETAILED DESCRIPTION:
The study was planned and conducted as a randomized controlled experiment. The sample of the randomized controlled trial consisted of 70 patients who applied to the emergency department with a migraine attack and met the study criteria. Data were collected via Patient Information Form, 24-Hour Migraine Quality of Life Scale, Visual Analogue Scale, Sphygmomanometer, and Pulse oximeter. Along with the medical treatment, patients of experimental group were massaged for 15 minutes with an aromatic oil mixture (lavender and peppermint) applied on the temple and root of the neck, and this application continued for three weeks. Control group patients, however, received only medical treatment. Descriptive statistics methods, Shapiro Wilks test, Wilcoxon Signed Ranks Test, Mann Whitney U Test, Kruskal Wallis Test, Fisher's Exact Test and Chi-Square Test were used for data evaluation.

ELIGIBILITY:
Inclusion Criteria:

diagnosed with migraine according to International Headache Society 2013 Being able to speak Turkish, being between the ages of 18 and 50, being literate, not having any communication problems, agreeing to participate in the study, having vital signs within normal limits not being diagnosed with a psychiatric disorder

Exclusion Criteria:

having a headache other than migraine being the ages under the 18 having any communication problems, having vital signs above or under normal limits being diagnosed with a psychiatric disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 83 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
24-Hour Migraine Quality of Life | After 30 minutes of medical treatment and massage, blood pressure, oxygen saturation and pain were reevaluated and "24-Hour Migraine Quality of Life Scale" was administered.
  The scale measures the change in quality of life for 24 hours after medication to relieve migraine headache.There are a total of 15 questions on the 7 Point Likert Scale. The scale has five domains for the quality of life, each with three items. These are migraine symptoms, emotions-concerns, work functioning, social functioning and energy-vitality.

IPD SHARING:
Plan to Share IPD: No